CLINICAL TRIAL: NCT07208877
Title: NTproBNP2 Test Kit (Time-Resolved Immunofluorescence Method) Clinical Evaluation Study Protocol
Brief Title: AQT90 FLEX NTproBNP (N-terminal Pro-brain Natriuretic Peptide) 2 Test Kit - Clinical Evaluation Study Protocol - China
Status: Not yet recruiting | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-092723
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Diagnostic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To validate the NTproBNP2 Test Kit by using the test results of the predicate device as a reference. It will be demonstrated that the investigational product (NTproBNP2 Test Kit) and the predicate are equivalent. Subsequently, it will be demonstrated that the investigational product can be used in clinical testing.

ELIGIBILITY:
Inclusion Criteria:

Samples that meet all the following criteria will be eligible for enrollment:

1. Samples from subjects with current or previous signs and/or symptoms of heart failure, or diagnosed heart failure.
2. Sample-related information is available, including a unique and traceable number, sample type, age, gender, date of sample collection, and clinical diagnosis, etc..
3. The sample volume is adequate, no less than 2 mL of whole blood.
4. The sample collection shall meet the informed consent waiver requirements of the ethics committee.

Exclusion Criteria:

Samples that meet any of the following criteria will be excluded:

1. Duplicate collection of samples from the same subject.
2. Samples that do not meet the collection, handling, and storage requirements outlined in the product's instructions for use.
3. Samples that are suspected of being poor quality, i.e. samples suspected of containing clots, visible hemolysis or lipids, or samples suspected of being contaminated with possible interfering substances.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study should select subjects that cover the intended population, considering differences in disease, age, and gender. It should not focus on a specific age group to ensure population representativeness. The samples (from the subject) contain interference also need to be involved.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
AQT90 FLEX NTproBNP2 Test Kit - Clinical Evaluation - China | 12 months
  Clinical evaluation indicator: The correlation coefficient between the investigational reagent and the predicate.
  Evaluation criteria: The correlation coefficient between the investigational reagent and the predicate shall not be less than 0.95. The slope should be within the range of [0.9, 1.1]. If this requirement is not met, it is recommended to increase the sample size and provide a detailed rationale.